CLINICAL TRIAL: NCT02917265
Title: Transcutaneous Vagus Nerve Stimulation for the Treatment of Systemic Lupus Erythematosus
Brief Title: Transcutaneous Vagus Nerve Stimulation for the Treatment of Lupus
Acronym: TRUST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Aikaterini Thanou (Individual)
Collaborators: Oklahoma Medical Research Foundation (Other); University of Oklahoma (Other)
Responsible Party: Principal Investigator, Aikaterini Thanou, Research Affiliate, Oklahoma Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H15-141
Record Dates: First submitted 2016-03-28; First posted 2016-09-28 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2019-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: vagus nerve stimulation; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TENS for vagus stimulation (Experimental): A transcutaneous electrical nerve stimulation (TENS) unit is applied to an area of the external ear that is innervated by the auricular branch of the vagus nerve.
  Interventions: Device: TENS for vagus stimulation
- TENS for sham stimulation (Sham Comparator): A TENS unit is applied to an area of the external ear that is devoid of vagus innervation.
  Interventions: Device: TENS for sham stimulation

INTERVENTIONS:
Device: TENS for vagus stimulation — TENS electrodes are applied on an area of the external ear innervated by the auricular branch of the vagus nerve.
  Arms: TENS for vagus stimulation
Device: TENS for sham stimulation — TENS electrodes are applied on an area of the external ear devoid of vagus innervation.
  Arms: TENS for sham stimulation

SUMMARY:
This is a 3-month double blinded randomized controlled study of transcutaneous electrical vagus nerve stimulation (tVNS) compared to a sham stimulation for the treatment of patients with active systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
Patients with SLE and active, non-organ-threatening disease are eligible to participate in this prospective randomized double blind trial of active or sham transcutaneous electrical vagus nerve stimulation (tVNS). Active tNVS is performed by the use of a transcutaneous electrical nerve stimulation (TENS) device with electrodes attached to an area of the external ear innervated by the auricular branch of the vagus nerve. The same protocol is followed in the sham tVNS arm, but the pads are placed on an area of the external ear that is devoid of vagus innervation.TENS is applied for 60 to 120 minutes daily as tolerated and participants keep a detailed log of their daily TENS sessions. Patients return to clinic at weeks 4, 8 and 12 for study related assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with SLE age 18-70 meeting the American College of Rheumatology Classification Criteria. Patients need to meet a minimum of 4 out of 11 criteria simultaneously or serially on two separate occasions.
2. Positive antinuclear antibody or anti-dsDNA within one year of screening
3. Non-serological SLEDAI ≥4 or ≥1 BILAG B or A and presence of inflammatory arthritis (defined by at least 3 swollen and 3 tender joints) at screening
4. Patients may receive on one or more of the following immune suppressive therapies: hydroxychloroquine, quinacrine, methotrexate, azathioprine, mycophenolate mofetil, tacrolimus, sirolimus, belimumab, abatacept. Immune suppressive medications should have been administered at stable doses for ≥30 days prior to baseline. Patients may also be on prednisone up to 10mg daily or equivalent steroid treatment at the baseline visit.

Exclusion Criteria:

1. Acute lupus nephritis defined as class II,III, IV or V nephritis diagnosed within 6 months or prot/creat > 1.5 gm/gm due to active lupus or in process of receiving induction therapy for nephritis
2. Active CNS lupus affecting mental status
3. Any other organ threatening or life threatening manifestation of SLE as well as those, who, in the opinion of the investigator, have severe multi-organ or refractory lupus
4. Rituximab treatment within 6 months prior to screening and/or without return of B cells to baseline levels
5. Treatment with cyclophosphamide within a month prior to screening
6. Treatment with any investigational drug within 3 months or 5 half-lives whichever is longer
7. Recurrent vaso-vagal syncopal episodes
8. Unilateral or bilateral vagotomy
9. Presence of any evidence of vagus nerve pathology or injury
10. Heart failure (NYHA class III or IV)
11. Known atherosclerotic disease, including severe carotid artery disease, uncontrolled hypertension, uncontrolled diabetes, and history of myocardial infarction (MI), cardiomyopathy or stroke within the past year. Clinically stable patients with coronary artery disease, but no recent MI (within the past year) and no current symptoms of angina are not however excluded.
12. Valvular and other structural heart disease that is evident by transthoracic echocardiogram and is associated with heart failure (NYHA class III or IV)
13. Prolonged QT interval or abnormal baseline ECG - sick sinus syndrome, Mobitz type 2 second or third degree heart block, atrial fibrillation, atrial flutter, recent history of ventricular tachycardia or ventricular fibrillation or clinically significant premature ventricular contraction
14. Individuals currently implanted with an electrical and/or neurostimulator device, such as cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant
15. Known respiratory disease that has decreased any pulmonary function test more than 25% below expected values or has resulted in hospitalization within the past year
16. All diagnosed syndromes affecting the central nervous system (CNS) or autonomic nervous system
17. Major psychiatric disorders including evidence of major depressive disorder (DSM-5 diagnostic criteria) that is not currently controlled by medications
18. Hemoglobin below 9.0 gm/dL (by the most recent CBC)
19. Pregnancy or breast feeding
20. Inability or unwillingness to understand and/or sign informed consent
21. Any other medical condition, whether or not related to lupus, which, in the opinion of the investigator, would render the patient inappropriate or too unstable to complete the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aikaterini Thanou, MD, Principal Investigator — Oklahoma Medical Research Foundation
Locations (1):
- Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Rheumatology Research Clinic of the Oklahoma Medical Research Foundation between 9.2015 and 5.2017.
Pre-assignment Details: Screening and randomization occurred at the same visit. One individual failed screening due to severe depression.
Groups:
- TENS for Vagus Stimulation: A transcutaneous electrical nerve stimulation (TENS) unit is applied to tragus, the area of the external ear innervated by the auricular branch of the vagus nerve.
  TENS for vagus stimulation: TENS electrodes are applied the tragus of the external ear.
- TENS for Sham Stimulation: A TENS unit is applied to the earlobe, an area of the external ear that is devoid of vagus innervation.
  TENS for sham stimulation: TENS electrodes are applied on the earlobe.
Period: Overall Study
Arm/Group | TENS for Vagus Stimulation | TENS for Sham Stimulation
Started (11.2015) | 5 | 2
Completed (5.2017) | 3 | 2
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TENS for Vagus Stimulation | TENS for Sham Stimulation | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 50 [25 to 69] | 51.5 [43 to 60] | 50.4 [25 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) [Mean (Full Range); unit: units on a scale] — The SLEDAI is the sum score of 24 variables to assess global lupus disease activity in the preceding 30 days. Scores can range from zero (no disease activity) to 105 (very active systemic lupus).
  Disease activity categories: no activity: SLEDAI = 0, mild disease activity: SLEDAI = 1-5, moderate disease activity: SLEDAI = 6-10, high disease activity: SLEDAI = 11-19, very high disease activity: SLEDAI >20
  units on a scale | 4.6 [4 to 6] | 4 [2 to 6] | 4.4 [2 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on Active vs Sham tVNS With Improvement in SLE Disease Activity by the BILAG-based Combined Lupus Assessment (BICLA)
Description: Achieving a BICLA response requires to meet all of the following parameters:
  1. All British Isles Lupus Assessment Group (BILAG) A scores improving to B/C/D and all BILAG level B scores improving to C/D
  2. No single new BILAG A & not >1 new BILAG B scores, no worsening of the baseline Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) total score AND no worsening in the Physician Global Assessment (PGA) (<10% worsening from baseline)
  3. No initiation of non-protocol treatments or premature study discontinuation
  The range of values for the above instruments are listed below, with higher scores indicating more active disease:
  BILAG: 0 to 96 SLEDAI: 0 to 105 PGA: 0-3
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TENS for Vagus Stimulation | TENS for Sham Stimulation
Number analyzed (Participants) | 5 | 2
Participants
  BICLA responders | 1 | 0
  BICLA non responders | 4 | 2
Statistical Analysis 1: Comparison: TENS for Vagus Stimulation vs TENS for Sham Stimulation; Test type: Superiority; p = 0.05, Chi-squared

2. Secondary Outcome: Percentage of Participants on Active vs Sham tVNS With Improvement in SLE Disease Activity by the Systemic Lupus Erythematosus Responder Index (SRI-4)
Description: SRI requires meeting all of the following parameters:
  1. ≥4-point reduction from baseline in the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score
  2. No single new British Isles Lupus Assessment Group (BILAG) A score & not >1 new BILAG B scores AND no worsening in the Physician Global Assessment (PGA) (<10% worsening from baseline)
  3. No initiation of non-protocol treatments or premature study discontinuation
  The range of values for the above instruments are listed below, with higher scores indicating more active disease:
  BILAG: 0 to 96 SLEDAI: 0 to 108 PGA: 0-3
Time Frame: 12 weeks
Population: all patients randomized to active treatment or placebo that had a total SLEDAI score of at least 4 at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | TENS for Vagus Stimulation | TENS for Sham Stimulation
Number analyzed (Participants) | 4 | 2
Participants
  SRI Responders | 0 | 0
  SRI Non-responders | 4 | 2

3. Secondary Outcome: Percentage of Participants on Active vs Sham tVNS With Improvement in Heart Rate Variability (HRV)
Description: HRV is measured by time domain (RMSSD and pNN50) and frequency domain [high frequency (HF), low to high frequency (LF/HF) ratio] parameters.
Time Frame: 12 weeks
Population: Analysis not done.
Arm/Group | TENS for Vagus Stimulation | TENS for Sham Stimulation
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Percentage of Participants on Active vs Sham tVNS That Experience an SLE Flare by SELENA SLEDAI Flare Index
Description: The SELENA SLEDAI flare index captures flares in the preceding 30 days by a combination of clinical descriptors and medications rules.
Time Frame: 12 weeks
Population: Analysis has not been done.
Arm/Group | TENS for Vagus Stimulation | TENS for Sham Stimulation
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Percentage of Participants on Active vs Sham tVNS With Improvement in Quality of Life Measured by the Lupus QoL
Description: The Lupus QoL is a patient reported outcome developed for measurement of quality of life of patients with SLE in clinical research
Time Frame: 12 weeks
Population: Analysis not done.
Arm/Group | TENS for Vagus Stimulation | TENS for Sham Stimulation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks (baseline to Month 3)
Arm/Group | TENS for Vagus Stimulation | TENS for Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 4/5 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TENS for Vagus Stimulation (N=5) | TENS for Sham Stimulation (N=2)
Urinary tract infections (Renal and urinary disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
paresthesias (Nervous system disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT02917265/Prot_SAP_001.pdf